CLINICAL TRIAL: NCT04572022
Title: Impact of Mobile Health Technology Application on Proximal Humerus Fracture Care Practice and Patient Self-Care Outcomes - A Pilot Randomized Controlled Trial
Brief Title: Impact of Mobile Health Technology Application on Proximal Humerus Fracture Care Practice
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Zehra Abdul Muhammad, Instructor (Research), Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5155
Record Dates: First submitted 2020-09-23; First posted 2020-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Proximal Humerus Fracture; Trauma
Keywords: Proximal Humerus Fracture; mobile Health application; rehabilitation exercises; patient teaching video modules
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups (intervention and control) in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group rehabilitation teaching video instructions (Experimental): Intervention group receive proximal humerus fracture standard care with additional mobile health shared step-wise rehabilitation teaching video instructions module.
  Interventions: Other: Step wise post-procedure mobile health shared rehabilitation teaching video instructions modules (as per fracture type)
- Control group (No Intervention): Control group receive proximal humerus fracture standard care only.

INTERVENTIONS:
Other: Step wise post-procedure mobile health shared rehabilitation teaching video instructions modules (as per fracture type) — Intervention group receive proximal humerus fracture standard care with additional mobile health shared step-wise rehabilitation teaching video instructions modules (as per fracture type). Classic Blue tooth technology will be utilized for teaching information sharing from doctor to the patient.
  Arms: Intervention group rehabilitation teaching video instructions

SUMMARY:
Proximal humerus fracture patient's upper limb complete function restoration mainly depends on patient rehabilitation exercises. One time teaching in clinic is usually not sufficient for patients to learn their rehabilitation exercises. This leads to delayed patient recovery and dis-satisfaction to treatment provided by health care providers.

Our aim is that mobile health technology might facilitate patient to easily access health related teaching information other than routine care to support patient in their self-health care management thus leading to proximal humerus fracture patient treatment outcome improvement.

Hypothesis:

Mobile health technology positively improves clinical and functional outcomes of proximal humerus fracture using validated outcome scoring scales.

Objectives:

Primary objective:

1. To improve adult proximal humerus fracture patient's clinical and functional outcomes using validated outcome scoring scales resulting in timely recovery with the help of patient self-health care capacity using mobile health app.
2. To compare patient clinical and functional outcomes by validated scoring scales between using mobile health app versus standard care.

Secondary Objective: To increase patient and doctor satisfaction rate in perspective with treatment provision usefully by digital technology application.

Methods:

Study design: Patient-centered, open labelled, parallel (1:1), pilot randomized controlled trial.

Total 60 subjects required with 30 in each arm in 24-month duration.

Study procedures:

1. Proximal humerus rehabilitation exercises video will be prepared after obtaining written informed consent from designated orthopaedic residents/surgeon.
2. Patients of 18 to 58 years of age with trauma associated proximal humerus fractures, who or their attendants are willing to participate. Patients who requires special care, patient not willing to exercise at home without physiotherapist support or participate in survey questionnaire and patients who does not have facility of classic blue tooth connectivity will be excluded.
3. Written informed consent will be administered the study subjects as per GCP guideline.
4. Each eligible patient will be randomized into intervention or control group.

   1. Intervention group: Classic Blue tooth technology will be utilized for interoperable solution of teaching video information sharing from doctor to patient. The end users will be enrolled trauma associated proximal humerus fracture patients whether treated surgically or conservatively.
   2. Control group: Routine care will be provided to control group and as per routine.
5. The patient will be followed at 6 weeks, 3 and 6 months. Data will be collected on Case report form by assigned person. Clinical and functional outcomes will be assessed by assigned person using Quick DASH and Oxford shoulder score.
6. Researchers will be trained on data collection form prior to data collection. In case of lost to follow-up, patients will be contacted by telephone.
7. Patient satisfaction questionnaire: Administered to intervention group only about impact of digital technology application on their health improvement and care outcomes.
8. Doctor satisfaction questionnaire: To assess treating surgeon satisfaction rate for digital technology application impact on intervention group patients' care and outcomes.
9. The research study does not seem to have any potential health hazard. As per Food and Drug Administration and GCP recommendations for Serious/Adverse event (SAE/AE), any patient who experience SAE/AE, will receive good clinical care at earliest and all relevant reporting bodies will be notified.
10. Data management will be carried out at the Department of Surgery. Subject data confidentiality will be maintained. After study completion, data will be archived and retained for maximum years.

Statistical Consideration:

Quantitative variables will be expressed as mean ± standard deviation and qualitative variables as frequencies (percentages). The efficacy on the basis of clinical and functional outcome and the AEs/SAEs will be assessed by intention to treat analysis. For group comparisons of clinical and functional categorical outcomes, chi-square test or Fisher Exact will be applied. p-values of less than 0.05 will be considered as statistically significant with a confidence interval of 95%.

Patient and doctor satisfaction scores will be analyzed using regression analysis. For Assessment of outcomes, repeated measure ANOVA and generalized estimating equation will be used. Multiple regression will be used to assess the association between multiple covariates.

DETAILED DESCRIPTION:
Due to complex anatomy with delayed recovery of proximal humerus fracture patients, there is high need of optimal treatment planning and care delivery process improvement to achieve better treatment outcomes. For current study, musculoskeletal service line at AKU will implement mobile health application specifically for proximal humerus trauma associated fracture patients which is simple to use. Internationally physiotherapy specialty related specific exercises are applied which is bit different from current study in the context of specialty and application. Mostly their focus is on rehabilitation of cases like scoliosis, dementia etc. This is the first time that orthopaedic specialty related, trauma associated, proximal humerus fracture specific modules will be developed with no advance IT based software application due to limited resources and to adhere to the patient data confidentiality. The application will be simple and user-friendly.

For current pilot trial research question is whether mobile health app. improve proximal humerus fracture patient treatment outcomes compared to standard care? Adhering to patient data confidentiality, our aim is that mobile health technology might facilitate patient to easily access health related teaching information other than routine care to support patient in their self-health care management thus leading to proximal humerus fracture patient treatment outcome improvement.

As proximal humerus fracture patient upper limb complete function restoration mainly depends on patient rehabilitation exercises, one time teaching in clinic by surgeons or physiotherapist is usually not sufficient for patients to learn their home rehabilitation exercises in routine practice. This leads to delayed patient recovery and dis-satisfaction to treatment provided by health care providers. Besides standard care, administering teaching video teaching modules with the help of mobile technology specifically for proximal humerus fracture patients might improve patient complete function restoration. Thus, mobile health strategy possibly will assist orthopaedic clinical team to reduce patient visit time, improve patient clinical and functional outcomes with increase in patient satisfaction and quick recovery.

Hypothesis:

Mobile health technology positively improves clinical and functional outcomes of proximal humerus fracture using validated outcome scoring scales.

Objectives:

1. Primary objective:

   1. To improve adult proximal humerus fracture patient's clinical and functional outcomes using validated outcome scoring scales resulting in timely recovery within four months post procedure with resumption of approximately 80% of patient upper limb function with the help of patient self-health care capacity using mobile health app.
   2. To compare patient clinical and functional outcomes by validated scoring scales between using mobile health app versus standard care.
2. Secondary Objective: To increase patient and doctor satisfaction rate in perspective with treatment provision usefully by digital technology application and health information sharing in health care settings.

Methods:

Number of participants:

The minimum sample size that investigator will require is 60 with 30 in intervention arm and 30 in control arm.

Study design: Patient-centered, open labelled, parallel (1:1), pilot randomized controlled trial. (Intervention group receive proximal humerus fracture care with mobile health shared rehabilitation teaching video instructions and control group will receive routine care for proximal humerus fracture as recommended by the treating surgeons).

Study Duration: 24 months

Study procedures: Study procedures will comply with all necessary ethical, Institutional and legal requirements.

1. In first step of the study, written informed consent will be obtained from designated orthopaedic residents/surgeon prior to video production. Proximal humerus rehabilitation exercises video will be prepared by orthopaedic resident or surgeon under observation of participating surgeon's expertise in which step wise rehabilitation exercises will be demonstrated exclusively for patient's teaching.
2. Patient eligibility criteria: Patients of 18 to 58 years of age with trauma associated proximal humerus fractures, presented at Orthopaedic inpatient and outpatient units, AKU who or their attendants are willing to follow the rehabilitation instructions via mobile application at home until completion of study follow up visits and agree to participate in very small survey questionnaire in the end of study will be selected. Patients who in special circumstances requiring special care and handling by expert health care providers, patient not willing to exercise at home without physiotherapist support or participate in survey questionnaire and patients who does not have facility of classic blue tooth connectivity for video download will be excluded.
3. Written informed consent will be administered by designated person as per good clinical practice guideline and obtained from the study subjects within the time of initial hospital arrival to follow-up within 21days post procedure.
4. Randomization: After obtaining written informed consent, on the same day, each eligible patient will be randomized into intervention or control group by randomly generated treatment allocation, sealed envelope technique will be used.

   1. Intervention group: Classic Blue tooth technology will be utilized for interoperable solution of teaching information sharing from doctor to patient. The end users will be enrolled trauma associated proximal humerus fracture patients whether treated surgically or conservatively. The video will be divided into 3 modules depending on proximal fracture type. Each module will reflect the necessary steps of exercises routinely taught by treating surgeons at clinics during subsequent follow-up visits. The rehabilitation video module (as per fracture type) will be transferred immediately at first post-procedure patient follow-up. For assessing patient compliance, it is routine care practice by orthopaedic surgeons to clinically judge patients for exercise adherence.
   2. Control group: Routine care will be provided to control group and as per routine.
5. Patient follow-ups and Data Collection: Patients will be followed at subsequent visits after treatment. The patient will be followed at 6±1 weeks, 3 months ±2 weeks and 6±1 months. Data will be collected on Case report form by assigned person. Clinical and functional outcomes will be assessed by assigned person using Quick DASH and Oxford shoulder score.
6. In order to reduce bias, researchers will be trained on data collection form prior to data collection. In case of lost to follow-up, patients will be contacted by telephone to gather necessary information.
7. Patient satisfaction questionnaire: At last follow-up, a small questionnaire by research team will be administered by assigned person to intervention group only about impact of digital technology application on their health improvement and care outcomes.
8. Doctor satisfaction questionnaire: A small questionnaire by research team will be administered to assess treating surgeon satisfaction rate for digital technology application impact on intervention group patients' care and outcomes.
9. The research study does not seem to have any potential health hazard. Complying with all regulatory standards and as per International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Good Clinical Practice (GCP) guidelines, study subjects will be provided optimum care at earliest.
10. As per Food and Drug Administration (FDA) and GCP definitions and recommendations for Serious/Adverse event (SAE/AE), any patient who experience SAE/AE, will receive good clinical care at earliest and all relevant reporting bodies will be notified. Designated research team member will be responsible to notify the SAE and AE timely to the Principal Investigator and prepare report with complete event details. Principal Investigator is responsible for sending reports to the reporting bodies (Ethical Review Committee, Sponsor etc.) as required, reviewing reports of adverse events (AEs) and serious adverse events (SAEs) that are submitted by designated research team member, identify safety concerns quickly and address in the report appropriately
11. Study Close-out: Study close-out process will be of two-month duration. Study progress report and all study closing steps will be carried out during this time with manuscript writing and study report submission.

Sampling Method: Non-probability, consecutive sampling

Data management Data management, randomization and the statistical analysis will be carried out at the Department of Surgery. Data entry will be conducted electronically and analyzed on SPSS version 19.0. Fifteen percent of the data will be double checked/validated by the Principal Investigator. Subject data confidentiality will be maintained by assigning subject ID, data entry by assigned person only on password protected system and keeping hard copies in lock and key. After study completion, data will be archived and retained for maximum years as recommended by Institutional and regulatory requirements.

Statistical Consideration:

The Statistical Package for Social Sciences (SPSS) version 19.0 will be used to analyze data. Quantitative variables will be expressed as mean ± standard deviation and qualitative variables as frequencies (percentages). The efficacy in intervention group on the basis of successful clinical and functional outcome achievement and the safety in intervention group on the basis of reported AEs/SAEs will be assessed by intention to treat analysis (ITT). The p-values for Group comparisons of clinical and functional categorical outcomes will be generated by chi-square test or Fisher Exact value of less than 0.05 will be considered as statistically significant with a confidence interval of 95%.

To patient and doctor satisfaction scores will be analyzed using regression analysis. For Assessment of outcomes at 6 weeks, 3 months and 6 months Investigator will use repeated measure ANOVA and generalized estimating equation (GEE). Multiple regression will be used to assess the association between multiple covariates and numeric outcome.

Device Safety:

No specific harm has been demonstrated by limited use of classic blue tooth technology up to date. Still if any adverse event is encountered like headache due to video based learning, increasing pain and/or numbness at the affected anatomical site, worsening range of motion etc., will be reported at the same time to the Institutional and other regulatory authorities as required and recommended by the Sponsor using telephone and e-mail. SAEs will be reported within 24 hours of knowing the event via telephone and e-mail. The completed forms will be submitted in time as recommended by the Sponsor otherwise within 10 days of knowing the event.

Withdrawals:

If patients would like to withdraw from the study due to any reason, he/she may stop participating in the research at any time without losing any of his/her patient rights. On the other hand, if in view of Principal Investigator, the subject is non-compliant and non-cooperative, he/she has right to withdraw the subject from the research study.

ELIGIBILITY:
Inclusion Criteria:

* Trauma associated proximal humerus fractures, presented at orthopaedic inpatient and outpatient units at Aga Khan University Hospital.
* Patient and/or their care providers are voluntarily willing to follow the rehabilitation instructions via mobile application at home until completion of study follow up visits.
* Patient agree to participate in very small survey questionnaire in the end of study.

Exclusion Criteria:

* Patients who in special circumstances requiring special care and handling by expert health care providers.
* Patient not willing to participate/exercise at home without physiotherapist support or to participate in survey questionnaire.
* Patients who does not have facility of classic blue tooth connectivity for video download.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Clinical and functional outcomes using validated outcome scoring scale | Four months after procedure with resumption of approximately 80% of patient upper limb function.
  Assessing improvement in proximal humerus fracture patient's clinical and functional outcomes using validated The Disabilities of the Arm, Shoulder and Hand Score (Quick DASH) with minimum to maximum score ranges from 0 (no disability) to 100 (severe disability) resulting in timely recovery with the help of patient self-health care capacity using mobile health app.
Clinical and functional outcomes using validated outcome scoring scale | Four months post procedure with resumption of approximately 80% of patient shoulder function.
  Assessing improvement in proximal humerus fracture patient's clinical and functional outcomes using validated Oxford shoulder score ranged from 0 (most impaired) to 48 (least impaired), resulting in timely recovery with the help of patient self-health care capacity using mobile health app.
Compare patient clinical and functional outcomes | 6 months
  Compare percentage of patients with clinical and functional outcomes improvement between mobile health app versus standard care by using Quick DASH score with interpretation of scores 0 to 24 is good, 25 to 49 is fair, 50 to 74 is poor and 75 to 100 is severe disability and by Oxford shoulder score with interpretation of scores 0 to 19 = Severe shoulder joint function, Score 20 to 29 = Moderate to severe shoulder joint function, Score 30 to 39 = Mild to moderate shoulder joint function, Score 40 to 48 = Satisfactory shoulder joint function.

SECONDARY OUTCOMES:
Patient and doctor satisfaction: rating | 6 months
  Patient and doctor satisfaction rate by using Patient Satisfaction Questionnaire and Doctor Satisfaction Questionnaire with minimum to maximum score ranges from 0 (strong disagreement with no satisfaction) to 25 (strong agreement with high satisfaction) in perspective with treatment provision usefully by digital technology application and health information sharing in health care settings.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra A Muhammad, M.B.B.S., MS, Principal Investigator — Aga Khan University Hospital, Karachi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual-patient data sharing of patient demographics, outcomes, SAE/AE.
  Study protocol (after study close-out) on request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Two years
Access Criteria: At the time of publication (deidentified individual patient data and analysis plan) and on request after study close-out (Study protocol, clinical study report).

REFERENCES:
- [Background] Dicianno BE, Parmanto B, Fairman AD, Crytzer TM, Yu DX, Pramana G, Coughenour D, Petrazzi AA. Perspectives on the evolution of mobile (mHealth) technologies and application to rehabilitation. Phys Ther. 2015 Mar;95(3):397-405. doi: 10.2522/ptj.20130534. Epub 2014 Jun 12. PMID 24925075
- [Background] Rehman H, Kamal AK, Sayani S, Morris PB, Merchant AT, Virani SS. Using Mobile Health (mHealth) Technology in the Management of Diabetes Mellitus, Physical Inactivity, and Smoking. Curr Atheroscler Rep. 2017 Apr;19(4):16. doi: 10.1007/s11883-017-0650-5. PMID 28243807
- [Background] Vriend I, Coehoorn I, Verhagen E. Implementation of an app-based neuromuscular training programme to prevent ankle sprains: a process evaluation using the RE-AIM Framework. Br J Sports Med. 2015 Apr;49(7):484-8. doi: 10.1136/bjsports-2013-092896. Epub 2014 Jan 27. PMID 24470587
- [Background] Milanese S, Gordon S, Buettner P, Flavell C, Ruston S, Coe D, O'Sullivan W, McCormack S. Reliability and concurrent validity of knee angle measurement: smart phone app versus universal goniometer used by experienced and novice clinicians. Man Ther. 2014 Dec;19(6):569-74. doi: 10.1016/j.math.2014.05.009. Epub 2014 Jun 4. PMID 24942491
- [Background] Yousaf K, Mehmood Z, Awan IA, Saba T, Alharbey R, Qadah T, Alrige MA. A comprehensive study of mobile-health based assistive technology for the healthcare of dementia and Alzheimer's disease (AD). Health Care Manag Sci. 2020 Jun;23(2):287-309. doi: 10.1007/s10729-019-09486-0. Epub 2019 Jun 20. PMID 31218511
- [Background] Laing BY, Mangione CM, Tseng CH, Leng M, Vaisberg E, Mahida M, Bholat M, Glazier E, Morisky DE, Bell DS. Effectiveness of a smartphone application for weight loss compared with usual care in overweight primary care patients: a randomized, controlled trial. Ann Intern Med. 2014 Nov 18;161(10 Suppl):S5-12. doi: 10.7326/M13-3005. PMID 25402403
- [Background] Zhang H, Jiang Y, Nguyen HD, Poo DC, Wang W. The effect of a smartphone-based coronary heart disease prevention (SBCHDP) programme on awareness and knowledge of CHD, stress, and cardiac-related lifestyle behaviours among the working population in Singapore: a pilot randomised controlled trial. Health Qual Life Outcomes. 2017 Mar 14;15(1):49. doi: 10.1186/s12955-017-0623-y. PMID 28288636
- [Background] Goyal S, Morita P, Lewis GF, Yu C, Seto E, Cafazzo JA. The Systematic Design of a Behavioural Mobile Health Application for the Self-Management of Type 2 Diabetes. Can J Diabetes. 2016 Feb;40(1):95-104. doi: 10.1016/j.jcjd.2015.06.007. Epub 2015 Oct 9. PMID 26455762
- [Background] Logan AG. Transforming hypertension management using mobile health technology for telemonitoring and self-care support. Can J Cardiol. 2013 May;29(5):579-85. doi: 10.1016/j.cjca.2013.02.024. PMID 23618506
- [Background] Mathews J, Lobenhoffer P. The Targon PH nail as an internal fixator for unstable fractures of the proximal humerus. Oper Orthop Traumatol. 2007 Aug;19(3):255-75. doi: 10.1007/s00064-007-1205-7. English, German. PMID 17728984
- [Background] Ye T, Wang L, Zhuang C, Wang Y, Zhang W, Qiu S. Functional outcomes following locking plate fixation of complex proximal humeral fractures. Orthopedics. 2013 Jun;36(6):e715-22. doi: 10.3928/01477447-20130523-14. PMID 23746032
- [Background] Zyto K. Non-operative treatment of comminuted fractures of the proximal humerus in elderly patients. Injury. 1998 Jun;29(5):349-52. doi: 10.1016/s0020-1383(97)00211-8. PMID 9813677